CLINICAL TRIAL: NCT05745649
Title: Restoration of Physical Function in Patients Following Total Knee Replacement: Comparison Between Resistive Strength Training Exercises & Ankle Weights
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 340
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A single blind RCT in which two groups were formulated. One as Control and other as an experimental
Who Masked: Participant
Masking Description: A single blind RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Resistive exercise
  Interventions: Other: Resistance exercises
- group B (Active Comparator): Ankle weights
  Interventions: Other: Ankle weights

INTERVENTIONS:
Other: Resistance exercises — Resistance exercises
  Arms: Group A
Other: Ankle weights — Ankle weights
  Arms: group B

SUMMARY:
Techniques used to restore the physical functions in TKR patients

DETAILED DESCRIPTION:
to restore the physical functions in TKR patients by the use of ankle weights and resistance exercises. Total 40 patients were included in this study and two groups had been formulated one as experimental and other as control. 2 sessions were given to each group for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients above 40 years with total knee arthroplasty
* 4-6 weeks following TKR

Exclusion Criteria:

* Age less than 40 patients
* Concurrent medical disease that could affect the progress (e.g., uncontrolled hypertension, advanced malignancy, decompensated cardiovascular disease.
* Pain score more than 6/10

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  zero means no pain and 10 means worst type of pain
Short form 36 Quality of life | 6 week
  on zero to 100 scale. minimum means low quality of life and higher values mean better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Rawal General & Dental Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided yet